CLINICAL TRIAL: NCT00465686
Title: Ergonomic Classroom Furniture and the Printing Legibility of Elementary School Students With CP
Brief Title: Effect of Ergonomic Classroom Furniture on the Printing Legibility of Elementary Students With Cerebral Palsy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Holland Bloorview Kids Rehabilitation Hospital (Other)
Responsible Party: Stephen Ryan, MSc, PEng/Scientist, Bloorview Research Institute, Bloorview Kids Rehab
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: 06-010
Record Dates: First submitted 2007-04-23; First posted 2007-04-25 (Estimated); Last update posted 2008-05-09 (Estimated); Status verified 2008-05

CONDITIONS: Cerebral Palsy
Keywords: handwriting; child; primary school; posture; assistive device
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Experimental)
  Interventions: Device: ergonomic chair and desk (Q-Learn Classic Chair and Q-Learn Desk); Device: ergonomic desk and chair (Q-Learn Desk)

INTERVENTIONS:
Device: ergonomic chair and desk (Q-Learn Classic Chair and Q-Learn Desk) — ergonomic school chair and desk adjusted to fit the child user as per the manufacturer's instructions
  Other Names: Q-Learn Classic Chair and Q-Learn Desk
Device: ergonomic desk and chair (Q-Learn Desk) — child sits on chair and desk for 5 minutes, then provides handwriting sample at one desk, then repeats this for the other desk
  Other Names: Q-Learn Desk

SUMMARY:
The purpose of this pilot study is to gather the data needed to do a larger research study to determine whether children with cerebral palsy print better sitting at an ergonomically-designed, custom-fitted school desk or at an oversized, standard school desk.

DETAILED DESCRIPTION:
This pilot study will allow us to gather information for a high-quality randomized controlled trial to study the efficacy of ergonomic school furniture as a remedial handwriting intervention for young students with cerebral palsy. We will conduct the study in two parts. In the first part, 30 children with Gross Motor Function Classification System (GMFCS) Level I and II cerebral palsy will each provide manuscript handwriting samples using two different school furniture configurations. A blinded assessor will score the legibility of handwriting samples using the Minnesota Handwriting Assessment (MHA) as a primary outcome measure. In the second part, seven occupational therapy experts will attend a focus group to help us determine the minimal clinically important difference score for the MHA. We will use the data collected to determine the sample size requirements for a proposed randomized controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* primary diagnosis of cerebral palsy
* functional status of Gross Motor Function Classification System Level I or II

Exclusion Criteria:

* genetic disorder;
* attention-deficit hyperactivity disorder; or,
* pervasive developmental disorder

Ages: 6 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2007-02; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
Minnesota Handwriting Assessment | 5-10 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Stephen E Ryan, MSc, PEng, Principal Investigator — Bloorview Research Institute, Bloorview Kids Rehab
Locations (1):
- Bloorview Research Institute, Bloorview Kids Rehab, Toronto, Ontario, Canada